CLINICAL TRIAL: NCT06837077
Title: A Single-center, Randomized, Crossover, Open-label Phase I Study to Compare the Safety and Pharmacokinetics of SHR-1209 Given as Single-site or Multiple-site Subcutaneous Injections in Healthy Volunteers
Brief Title: Study of SHR-1209 Administered by Single-site or Multiple-site Subcutaneous Injections in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1209-105
Record Dates: First submitted 2025-01-07; First posted 2025-02-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hypercholesterolemia and Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1209 single-site subcutaneous injection; Drug: SHR-1209 multiple-site subcutaneous injections
- Treatment group B (Experimental)
  Interventions: Drug: SHR-1209 single-site subcutaneous injection; Drug: SHR-1209 multiple-site subcutaneous injections

INTERVENTIONS:
Drug: SHR-1209 single-site subcutaneous injection — SHR-1209 single-site subcutaneous injection.
Drug: SHR-1209 multiple-site subcutaneous injections — SHR-1209 multiple-site subcutaneous injections.

SUMMARY:
In order to improve the medication convenience and compliance of patients and facilitates in the long-term control of disease condition, it is planned to reduced the number of injections to one per administration. The study aims to compare the safety and pharmacokinetics data to assess feasibility of single-site and multiple-site injection for administration.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the research procedures and methods, being able to complete the research in accordance with the procedure requirements, and sign the informed consent;
2. The age on the date of signing the informed consent must be ≥18 years old and ≤55 years old;
3. Body mass index (BMI) at screening period must be ≥19.0 kg/m2 and <28.0 kg/m2, weight of male must≥ 50.0 kg and <90.0 kg, and female≥ 45.0 kg and <90.0 kg;
4. The subjects and their female partners are willing to have no reproductive plan from signing the informed consent to 16 weeks after the last administration of the study drug, and voluntarily take effective contraceptive measures and do not plan to donate sperm or ovum.

Exclusion Criteria:

1. Serious infection within 3 months before screening;
2. History of food or drug allergy or atopic allergic disease (asthma, urticaria);
3. Positive blood pregnancy test;
4. Have a history of drug abuse;
5. Women who are pregnant or breastfeeding;
6. Subjects who are considered by the investigator to have any other factors which are not suitable for participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) was used to evaluate the injection site pain of single-site subcutaneous injection of SHR-1209. | After injection in day 1 and day 57.
Visual Analog Scale (VAS) was used to evaluate the injection site pain of multiple-site subcutaneous injections of SHR-1209. | After injections in day 1 and day 57.
Area under the curve (AUC0-56). | After injection in day 1 up to day 56.
Peak time (Tmax) of SHR-1209. | After injection in day 1 up to day 56.
Peak concentration (Cmax) of SHR-1209. | After injection in day 1 up to day 56.

SECONDARY OUTCOMES:
Subjects' preferred method of SHR-1209 administration between the tested injection regimens. | Day 68.
Incidence and severity of adverse events (AEs). | From Day 1 to Day 169.
Incidence and severity of serious adverse events (SAEs). | From Day 1 to Day 169.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided